CLINICAL TRIAL: NCT04132960
Title: Phase II, Open Label Study of DS-8201a, an Anti-HER2-antibody Drug Conjugate (ADC) for Advanced Breast Cancer Patients, With Biomarkers Analysis to Characterize Response/Resistance to Therapy
Brief Title: Study of DS-8201a, an Antibody Drug Conjugate for Advanced Breast Cancer Patients, With Biomarkers Analysis
Acronym: DAISY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-0105/1815; 2018-004868-57 (EudraCT Number)
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Breast Tumors
Keywords: DS-8201a; ADC; HER2; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Intervention Model Description: The main objective is to evaluate the anti-tumor activity of DS-8201a in three cohorts of advanced breast cancer patients:
  * Cohort 1: HER2 over-expressing (HER2 IHC3+ or HER2 IHC2+/ISH+)
  * Cohort 2: HER2 low-expressing (IHC1+ or IHC2+/ISH-)
  * Cohort 3: HER2 non-expressing (IHC0+)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HER2 status (Experimental): Three cohorts of advanced breast cancer patients:
  * Cohort 1: HER2 over-expressing (HER2 IHC3+ or HER2 IHC2+/ISH+)
  * Cohort 2: HER2 low-expressing (IHC1+ or IHC2+/ISH-)
  * Cohort 3: HER2 non-expressing (IHC0+)
  Interventions: Drug: DS-8201a

INTERVENTIONS:
Drug: DS-8201a — Anti-HER2-antibody drug conjugate (ADC)

SUMMARY:
Multicenter, open-label phase II trial assessing the efficacy of DS-8201a monotherapy in patients with metastatic breast cancer.

DETAILED DESCRIPTION:
The main objective is to evaluate the anti-tumor activity of DS-8201a in three cohorts of advanced breast cancer patients:

* Cohort 1: HER2 over-expressing (HER2 IHC3+ or HER2 IHC2+/ISH+)
* Cohort 2: HER2 low-expressing (IHC1+ or IHC2+/ISH-)
* Cohort 3: HER2 non-expressing (IHC0+)

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed a written informed consent form prior to any study specific procedures. When the patient is physically unable to give his/her written consent, a trusted person of his/her choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent.
2. Female or male subjects aged ≥18 years.
3. Patient with histologically-confirmed diagnosis of invasive breast cancer. Tumors can be either HER2 immunohistochemistry (IHC)3+/in situ hybridization (ISH) positive or IHC2+/ISH positive or IHC2+/ISH negative or IHC1+ or IHC0+, of most recent tumor tissue sample available.
4. Patient with a documented radiologic metastatic progression.
5. Patient considered by the investigator as not amenable to any other validated therapeutic option, after at least 1 line of chemotherapy in metastatic setting. Patient must have been previously treated with anthracyclines and taxanes (in (neo-)adjuvant and/or metastatic setting). Additionally:

   * Patient with HER2 over-expressing (IHC3+ and IHC2+/ISH+) tumor must have been treated and have progressed on trastuzumab and on TDM-1. Prior treatment with pertuzumab is not required.
   * Patient with HER2 negative (IHC0, 1+, and 2+/ISH-) and hormone receptor positive (estrogen receptor (ER)+ and/or progesterone receptor (PR)+) tumor must be resistant to endocrine therapy and CDK4/6 inhibitors, and must have been treated with capecitabine.
6. Non-bone metastatic site easily accessible to biopsy.
7. Presence of at least one measurable lesion according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
8. Patient with world health organization (WHO) performance status ≤1.
9. Adequate bone marrow function: absolute neutrophil count (ANC) ≥1.5 × 10⁹/L, platelet count ≥100 × 10⁹/L, and hemoglobin ≥9 g/dL (transfusion is not allowed within 1 week prior to baseline assessment).
10. Adequate liver function: total bilirubin level ≤1.5 × the upper limit of normal (ULN) range if no liver metastases or <3 x ULN in the presence of documented Gilbert's Syndrome or liver metastases. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤3 × ULN (AST and ALT≤ 5 ULN when documented liver metastasis).
11. Adequate blood clotting function: International Normalized Ratio (INR)/Prothrombin Time (PT) and activated Partial Thromboplastin Time (aPTT) ≤1.5 x ULN.
12. Adequate renal function: estimated creatinine clearance ≥30 mL/min according to the Cockcroft-Gault formula or serum creatinine ≤1.5 x ULN.
13. Adequate cardiac function: left ventricular ejection fraction (LVEF) ≥ 50% at baseline as determined by either echocardiogram (ECHO) or multigated acquisition (MUGA) scan within 28 days before inclusion.
14. Male and female subjects of reproductive/childbearing potential must agree to use of a highly effective contraception for subjects throughout the study and for at least 4.5 months after last study treatment administration if the risk of conception exists.
15. Women of childbearing potential must have a negative serum pregnancy test within 14 days of enrolment or urine pregnancy test 72 hours prior to enrolment.
16. Patient is willing to comply with 2 sequential tumor biopsies (baseline and at first progression), and with a series of blood samples throughout the study.
17. Patients must be affiliated to a Social Security System.

Exclusion Criteria:

1. Patient with a breast cancer amenable for resection or radiation therapy with curative intent.
2. Patient has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Subjects with clinically inactive brain metastases may be included in the study. Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy.
3. Patient with bone metastatic disease only.
4. Patient with multiple primary malignancies within 3 years, except adequately resected non-melanoma skin cancer, curatively treated in-situ disease, other solid tumors curatively treated, or contralateral breast cancer.
5. Persistent unresolved toxicities with grade ≥2 (except alopecia and renal function). Subject with chronic Grade 2 toxicities may be eligible per the discretion of the Investigator after consultation with the Sponsor (eg, Grade 2 chemotherapy-induced neuropathy).
6. Patient receiving treatments such as chemotherapy (including antibody drug therapy, retinoid therapy, hormonal therapy) within 3 weeks before inclusion (within 2 weeks or 5 half-lives, whichever is longer, for small-molecule targeted agents, within 6 weeks for nitrosureas or mitomycin C), immunotherapy within 4 weeks before inclusion, radiotherapy within 4 weeks (if palliative stereotactic radiotherapy: within 2 weeks) or major surgery within 4 weeks. Participation in other studies involving investigational drug(s) within 4 weeks prior to study entry and/or during study participation.
7. Patient using drugs that could have pharmacokinetics interaction with investigational drugs. Concomitant use of strong CYP3A4 inhibitors or OATP 1B inhibitors should be avoided. If concomitant use of strong CYP3A4 or OATP 1B inhibitors is unavoidable, consider delaying DS-8201a treatment until the inhibitors have cleared from the circulation (approximately 3 elimination half-lives of the inhibitors) when possible. If a strong CYP3A4 inhibitor or an OATP 1B inhibitor is co-administered and DS-8201a treatment cannot be delayed, patients should be closely monitored for adverse reactions.
8. Patients with a concomitant use of chronic systemic (intravenous or oral) corticosteroids or other immunosuppressive medications except for managing adverse events (inhaled steroids or intra articular steroid injections are permitted in this study.) Subjects with bronchopulmonary disorders who require intermittent use of bronchodilators (such as albuterol) will not be excluded from this study.
9. Patient with history of (noninfectious) interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
10. Patient with clinically significant corneal disease in the opinion of the Investigator.
11. Known prior severe hypersensitivity to investigational product or any component in its formulation, including known severe hypersensitivity reactions to study drug (National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 Grade ≥3).
12. Patient has a history of severe hypersensitivity reactions to other monoclonal antibodies.
13. Patients previously treated with topoisomerase 1 inhibitor.
14. Patient has substance abuse or any other medical conditions that would increase the safety risk to the subject or interfere with participation of the subject or evaluation of the clinical study in the opinion of the Investigator.
15. Known history of testing positive for HIV or known acquired immunodeficiency syndrome.
16. Known active hepatitis B virus or hepatitis C virus infection at screening.
17. Active infection requiring systemic therapy (as intravenous antibiotics, antivirals, antifungals,…).
18. Other severe acute or chronic medical conditions or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
19. Patient with a history of symptomatic congestive heart failure (New York Heart Association Class II to IV), serious cardiac arrhythmia requiring treatment, history of myocardial infarction or troponin levels consistent with myocardial infarction 28 days prior to inclusion, or unstable angina within 6 months prior to inclusion, or current dyspnea at rest due to advanced malignancy.
20. Patient with a corrected QT interval (QTc) prolongation to >470 ms (females) or >450 ms (males) based on average of the screening triplicate12-lead electrocardiogram (ECG).
21. Pregnant women, women who are likely to become pregnant or are breastfeeding or women who want donate, or retrieve for their own use, ova from the time of screening and throughout the study and for at least 4.5 months after last study treatment administration.
22. Patient with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
23. Patient unwilling to participate to the biological investigations.
24. Individual deprived of liberty or placed under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Antitumor activity of DS-8201a in the 3 cohorts of patients | 12 months
  The primary endpoint is antitumor activity of DS-8201a carried out by the determination of the confirmed best objective response (BOR) rate in each cohort. The BOR is defined as the presence of a confirmed partial or complete response observed on treatment, as assessed by investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique DIERAS, Principal Investigator — Centre Eugène Marquis
Locations (15):
- France (15):
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Universitaire Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Institut Curie - Hôpital Huguenin, Saint-Cloud
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Institut de Cancérologie Strasbourg Europe (ICANS), Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Mosele F, Deluche E, Lusque A, Le Bescond L, Filleron T, Pradat Y, Ducoulombier A, Pistilli B, Bachelot T, Viret F, Levy C, Signolle N, Alfaro A, Tran DTN, Garberis IJ, Talbot H, Christodoulidis S, Vakalopoulou M, Droin N, Stourm A, Kobayashi M, Kakegawa T, Lacroix L, Saulnier P, Job B, Deloger M, Jimenez M, Mahier C, Baris V, Laplante P, Kannouche P, Marty V, Lacroix-Triki M, Dieras V, Andre F. Trastuzumab deruxtecan in metastatic breast cancer with variable HER2 expression: the phase 2 DAISY trial. Nat Med. 2023 Aug;29(8):2110-2120. doi: 10.1038/s41591-023-02478-2. Epub 2023 Jul 24. PMID 37488289